CLINICAL TRIAL: NCT04677335
Title: Effect of a Nutritional Supplement (AB-LIFE Plus Monacolin K) to Reduce Total and LDL Cholesterol Levels
Brief Title: Combination of AB-LIFE Probiotic Plus Monacolin K to Reduce Blood Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: University of Extremadura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRIMACOL01
Record Dates: First submitted 2020-11-27; First posted 2020-12-21 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hypercholesterolemia
Keywords: Probiotic; Lactobacillus; Monacolin K; Monascus purpureus
MeSH Terms: conditions — Hypercholesterolemia | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceutical (Experimental): Nutraceutical capsules taken once daily for 12 weeks
  Interventions: Dietary Supplement: AB-LIFE with Monacolin K
- Control (Placebo Comparator): Placebo capsules taken once daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AB-LIFE with Monacolin K — Red yeast rice extract (also known by its scientific name, Monascus purpureus) certified to contain 10 mg of monacolin K, plus 1 billion total cfu of AB-LIFE probiotic formula, which is composed of 3 Lactoplantibacillus plantarum (formerly known as Lactobacillus plantarum) strains: CECT7527 (also known as KABP011™), CECT7528 (also known as KABP012™) and CECT7529 (also known as KABP013™), all in a maltodextrin carrier. Capsules are of vegetable origin (hydroxypropylmethyl cellulose).
  Arms: Nutraceutical
Other: Placebo — Placebo capsules containing maltodextrin carrier only. Capsules are of vegetable origin (hydroxypropylmethyl cellulose).
  Arms: Control

SUMMARY:
This randomized study evaluates the effectiveness of a nutraceutical combining billion colony forming units (cfu) of three L. plantarum strains (CECT7527, CECT7528 and CECT7529) and 10 mg of monacolin K in reducing blood cholesterol.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) are the number 1 cause of death globally, and retention of low-density lipoprotein cholesterol (LDL-C) and similar cholesterol-rich lipoproteins containing apolipoprotein B (ApoB) within the arterial wall is a key initiating event in CVDs. Statins are the mainstay of pharmacological cholesterol-reduction therapy. However, a significant proportion of patients report some degree of statin intolerance, which typically fade away when the statin is switched, discontinued or the dosage reduced. A growing attention has been devoted to the correction of increased LDL-C levels through the use of dietary supplements, either because some patients have milder forms of hypercholesterolemia or as an alternative to statins in patients who may have experienced or are worried of side effects. Nutraceutical combinations are increasingly used in clinical practice. In this pilot randomized study, we sought to evaluate of the effect on LDL-C and other blood lipid parameters of a nutraceutical combining Red Yeast Rice extract (also known by its scientific name Monascus purpureus) containing 10 mg of monacolin K, plus 1 billion colony forming units (cfu) of the AB-LIFE probiotic formula. The later is composed of three L. plantarum strains, namely CECT7527 (also known as KABP011™), CECT7528 (also known as KABP012™) and CECT7529 (also known as KABP013™).

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol (TC) ≥200 mg/dL and statin-naïve or having recently stopped statin treatment because of statin intolerance.

Exclusion Criteria:

* History of cardiovascular events or alcohol abuse, presence of diabetes, chronic advanced kidney disease, thyroid disorders, hepatic disorders, familial hypercholesterolemia or immunosuppression
* Body mass index (BMI) ≤ 18.5 or ≥40 Kg/m2
* Use of antibiotics within 4 weeks of study initiation, current use of other probiotics, lipid-lowering medications, corticoids, beta-blockers or calcium channel blockers, thiazide diuretics, estrogen replacement therapy
* Pregnant or lactating women
* Patients with other severe disease that could interfere with the results of the study.
* Patients not agreeing to maintain their usual physical activity throughout the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Change in low density lipoprotein cholesterol (LDL-C) | 0, 6 and 12 weeks
  Fasting serum levels of low density lipoprotein cholesterol (LDL-C), assessed by repeated measures analysis at three timepoints (baseline, mid of intervention and end of intervention).

SECONDARY OUTCOMES:
Change in total cholesterol (TC) | 0, 6 and 12 weeks
  Fasting serum levels of total cholesterol (TC), assessed by repeated measures analysis at three timepoints (baseline, mid of intervention and end of intervention).
Change in high density lipoprotein cholesterol (HDL-C) | 0, 6 and 12 weeks
  Fasting serum levels of high density lipoprotein cholesterol (HDL-C), assessed by repeated measures analysis at three timepoints (baseline, mid of intervention and end of intervention).
Change in triglycerides (TG) | 0, 6 and 12 weeks
  Fasting serum levels of triglycerides (TG), assessed by repeated measures analysis at three timepoints (baseline, mid of intervention and end of intervention).
Change in Body Mass Index (BMI) | 0 and 12 weeks
  Body Mass Index, calculated as body weight (in kilograms) divided by squared height (in meters), assessed by repeated measures analysis at two timepoints (baseline and end of intervention).
Change in body weight | 0 and 12 weeks
  Body weight in kilograms, assessed by repeated measures analysis at two timepoints (baseline and end of intervention).
Change in percent body fat | 0 and 12 weeks
  Percent of body fat (as determined with a MC780 Body Analyzer), assessed by repeated measures analysis at two timepoints (baseline and end of intervention).
Patient satisfaction with treatment | 12 weeks
  Rated with a Likert-type scale ranging 0 (very dissatisfied) to 4 (very satisfied), assessed at the end of the intervention.
Treatment-emergent adverse effects | 12 weeks
  Incidence of adverse effects (type and number) and relatedness to study product (using a 5 category system: certain, likely related, possibly related, conditionally related, unknown), as documented according to the Spanish Medicine and Medical Device Agency (AEMPS) pharmacovigilance system

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Guerrero Bonmatty, PhD, Principal Investigator — University of Extremadura (SPAIN)

IPD SHARING:
Plan to Share IPD: No